CLINICAL TRIAL: NCT04180930
Title: Psychometric Evaluation of the Clinician Administered PTSD Scale for DSM-5 (CAPS-5) and the PTSD Symptom Scale Interview for DSM-5 (PSSI-5) in an Active Duty and Military Veteran Sample
Brief Title: An Evaluation of Two PTSD Assessments in an Active Duty and Military Veteran Sample
Status: Recruiting | Type: Observational
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2017-7745
Record Dates: First submitted 2019-06-25; First posted 2019-11-29 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Assessment; Post-Traumatic Stress Disorder; PTSD; Veterans; Military
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood; saliva; PAXgene RNA; plasma; serum; buffy coat (optional)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: Individuals randomized to Cohort 1 will be assigned to the CAPS-5 and will complete between two and seven research visits. Participants will be administered the CAPS-5 during visit 2, and then will be randomized a second time into groups 1-A and 1-B. Group 1-A will end participation after visit 2. Group 1-B will complete visits 3-7 and will be administered the CAPS-5 at each of these visits along with other measures of cognitive and behavioral functioning, and will provide biofluid samples.
  Interventions: Diagnostic Test: CAPS-5
- Cohort 2: Individuals randomized to Cohort 2 will be assigned to the PSSI-5 and will complete between two and seven research visits. Participants will be administered the PSSI-5 during visit 2, and then will be randomized a second time into groups 2-A and 2-B. Group 2-A will end participation after visit 2. Group 2-B will complete visits 3-7 and will be administered the PSSI-5 at each of these visits along with other measures of cognitive and behavioral functioning, and will provide biofluid samples.
  Interventions: Diagnostic Test: PSSI-5
- Cohort 3: Individuals randomized to Cohort 3 will have three office visits and will complete the CAPS-5 and the PSSI-5 in a counter-balanced order during visits 2 and 3, along with other measures of cognitive and behavioral functioning, and will provide biofluid samples.
  Interventions: Diagnostic Test: CAPS-5; Diagnostic Test: PSSI-5
- Cohort 4: Individuals randomized to Cohort 4 will have three office visits and will complete the CAPS-IV and the CAPS-5 in a counter-balanced order during visits 2 and 3, along with other measures of cognitive and behavioral functioning, and will provide biofluid samples.
  Interventions: Diagnostic Test: CAPS-5; Diagnostic Test: CAPS-IV

INTERVENTIONS:
Diagnostic Test: CAPS-5 — Clinician Administered PTSD Scale for DMS-5
  Groups: Cohort 1; Cohort 3; Cohort 4
Diagnostic Test: PSSI-5 — PTSD Symptom Scale Interview for DSM-5
  Groups: Cohort 2; Cohort 3
Diagnostic Test: CAPS-IV — Clinician Administered PTSD Scale for DSM-IV
  Groups: Cohort 4

SUMMARY:
Given the high prevalence of post-traumatic stress disorder (PTSD) in veterans and active duty military, the focus of this research study is to test the reliability of two new PTSD assessments, the Clinician Administered PTSD Scale for DSM-5 (CAPS-5) and the PTSD Symptom Scale Interview for DSM-5 (PSSI-5) and compare the results between the two new assessments and the previous "gold standard", the Clinician Administered PTSD Scale for DSM-IV (CAPS-IV). Biomarkers believed to be related to PTSD (e.g., biofluid biomarkers, cognitive and physiological markers, and neural activity as measured by EEG) will be collected to inform targeted interventions in specific groups of patients and other large-scale biomarker discovery efforts in the field. Participants will be 950 male and female active duty military and veterans ages 18 or older who have been exposed to at least one traumatic event.

DETAILED DESCRIPTION:
This is a randomized, observational study where participants will be randomized into one of the four study cohorts. The primary goals of this study are to establish the test-retest reliability of the CAPS-5 and the PSSI-5 and to compare these with each other (Cohorts 1 and 2), to test the convergent validity of the CAPS-5 against the PSSI (Cohort 3) and against the CAPS-IV (Cohort 4), and finally to investigate the consistency of response over 12 weeks on CAPS-5 (Cohort 1) and on the PSSI-5 (Cohort 2). In addition, on an exploratory level, possible biomarkers of PTSD and their relationship to each other and to diagnosis of PTSD will be evaluated.

Participants will be 950 males and females recruited from the Cincinnati VA Medical Center (Cincinnati, OH), Trauma Recovery Center, and Tripler Army Medical Center (Honolulu, HI).

the investigators anticipate that understanding the validity and reliability of the PSSI-5 and the CAPS-5 and the biomarkers related to PTSD will provide necessary information for care provided to active duty military and veterans suffering from PTSD. It will also directly inform trial designs and increase the likelihood of technical and regulatory success for new treatments for PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female active duty personnel or military veterans, 18 years of age or older
* Competent to give informed consent
* Have experienced any Criterion A qualifying traumatic event as defined by the Life Events Checklist for DSM-5 (LEC-5)
* Score a 3 or above on the Primary Care-Post Traumatic Stress Disorder Screen (PC-PTSD-5)

Exclusion Criteria:

* Current suicidal or homicidal ideation with a plan, and substance use disorder requiring detoxification currently or in the past month as assessed using the SCID and Suicidal Ideation/Homicidal Ideation screening tool (SI/HI screen)
* Assessment using CAPS or PSSI in the previous 1 year
* Currently receiving psychotherapy or counseling for PTSD
* Moderate to sever cognitive impairment as measured by the Montreal Cognitive Assessment (MoCA)
* Meet criteria for unmedicated Bipolar I, Bipolar II, Schizophrenia, or other psychotic disorders in the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Active duty military personnel and veterans who satisfy the enrollment criteria. Study participants will be active duty personnel or veterans with PTSD symptoms, who may or may not meet diagnostic criteria for PTSD, recruit from up to two military treatment facilities (MTFs) and one VA facility.
Sampling Method: Non-Probability Sample
Enrollment: 950 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Test-Retest reliability of Clinician Administered PTSD Scale for DSM-5 (CAPS-5) Total Score | 7 days (+/- 2) between measurements
  Concordance of the Clinician Administered PTSD Scale Total Score of at 2 visits. The severity of diagnosed PTSD is determined by the total score. (minimum score of 0 = absent to a maximum score of 80 = extreme)
Test-retest reliability of PTSD Symptom Scale - Interview for DSM-5 (PSSI-5) Total Score | 7 days (+/- 2) between measurements
  To determine the test-retest reliability of Posttraumatic Stress Disorder Symptom Scale Interview-5 within Visits 2-3 for Groups 1-B and 2-B. The severity of diagnosed PTSD is determined by the total score. (minimum score of 0 = absent to a maximum score of 80 = extreme)
Correlation among the total scores of the CAPS-5, PSSI-5, and Clinician Administered PTSD Scale for DSM-IV (CAPS-IV) | Up to 39 days from the eligibility screen for Cohorts 1-4
  Correlation coefficient among the totals scores for 3 different PTSD symptom scales
Stability of the Clinician Administered PTSD Scale for DSM-5 (CAPS-5) item-level scores over 6 weeks | Up to 6 weeks for Group 1-B
  Change in the DSM-5 Clinician Administered PTSD Scale item-level scores over 6 weeks. The severity of diagnosed PTSD is determined by the total score. (minimum score of 0 = absent to a maximum score of 80 = extreme)
Stability of PTSD Symptom Scale - Interview for DSM-5 (PSSI-5) item-level scores over 6 weeks | Up to 6 weeks for Group 2-B
  Change in PTSD Symptom Scale for DSM-5 Posttraumatic Stress Disorder Symptom Scale Interview item-level scores over 6 weeks. The severity of diagnosed PTSD is determined by the total score. (minimum score of 0 = absent to a maximum score of 80 = extreme)

SECONDARY OUTCOMES:
Concordance rate between diagnostic tests | 7 days (+/- 2) between measurements
  To determine the concordance rate between diagnosis of PTSD using the CAPS-IV and CAPS-5, and the CAPS-5 and PSSI-5. The severity of diagnosed PTSD is determined by the total score. (minimum score of 0 = absent to a maximum score of 80 = extreme)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Chard, PhD, Principal Investigator — Cincinnati VA Medical Center, University of Cincinnati; Brian Marx, PhD, Principal Investigator — National Center for PTSD at VA Boston Healthcare System
Locations (3):
- United States (3):
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Cincinnati VA Medical Center - Trauma Recovery Center, Fort Thomas, Kentucky
  - Walter Reed National Military Medical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Final data sets resulting from this study will be shared outside the study team in de-identified format only. Data will be shared with study collaborators from the following institutions: VA Boston healthcare System, Stanford University, Palo Alto VA Health Care System, Auburn University, and the University of Pennsylvania. Research proposals from other institutions will be reviewed by a group of experienced scientists who will judge each request for its scientific merit, its potential contribution to the understanding of the disease, and for the qualifications of the research team. All data will be identified by a code number.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Starting in March 2020
Access Criteria: De-identified, anonymized databases will be shared electronically through the VA network and secure messaging. Only de-identified data will be made available outside the VA. The optional biofluid collection for future exploratory research will only be made available to investigators in a de-identified format with the permission of the sponsor, proper protocol approval, and human participants' protection in place.